CLINICAL TRIAL: NCT06397339
Title: Indian Transforming Alzheimer's Care Training (INTACT)
Acronym: INTACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: University of Washington (Other); University of Miami (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Patrik Johansson, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19630
Record Dates: First submitted 2024-03-15; First posted 2024-05-02 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
Keywords: ADRD, MCI
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Group Randomized Trial with 28 urban and rural clinics that serve AI/ANs in 11 states. INTACT will be randomized at the clinic level and delivered to PCPs in clinics. Most outcome data will be derived from EHRs and PCP surveys. The study will use an immediate intervention and waitlist control randomization pattern with clinics randomized to the immediate intervention group receiving the INTACT program after the baseline data collection and the waitlist control group after the 12-month follow-up data collection is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The INTACT Program has three components:
  1. provide a training for Primary Care Providers (PCPs) training in screening, diagnosis, and care for ADRD,
  2. at the PCP level, provide quarterly webinars. Topics will address driving and dementia; communication tips for someone with dementia; eating and drinking in advanced dementia; and advanced care planning for dementia.
  3. At the clinic level, provide a workflow model for cognitive evaluation and setting a plan for the newly diagnosed patient. The INTACT intervention lasts 12 months and Continuing Medical Education credits will be available to PCPs who complete the INTACT training program
  Interventions: Other: INTACT Program
- Waitlist (Other): The INTACT Program has three components:
  1. provide a training for Primary Care Providers (PCPs) training in screening, diagnosis, and care for ADRD,
  2. at the PCP level, provide quarterly webinars. Topics will address driving and dementia; communication tips for someone with dementia; eating and drinking in advanced dementia; and advanced care planning for dementia.
  3. At the clinic level, provide a workflow model for cognitive evaluation and setting a plan for the newly diagnosed patient. The INTACT intervention lasts 12 months and Continuing Medical Education credits will be available to PCPs who complete the INTACT training program
  Interventions: Other: INTACT Program

INTERVENTIONS:
Other: INTACT Program — The INTACT Program has three components:
  1. provide a training for Primary Care Providers (PCPs) training in screening, diagnosis, and care for ADRD,
  2. at the PCP level, provide quarterly webinars. Topics will address driving and dementia; communication tips for someone with dementia; eating and drinking in advanced dementia; and advanced care planning for dementia.
  3. At the clinic level, provide a workflow model for cognitive evaluation and setting a plan for the newly diagnosed patient. The INTACT intervention lasts 12 months and Continuing Medical Education credits will be available to PCPs who complete the INTACT training program

SUMMARY:
INTACT will utilize a group-randomized trial, to test the effectiveness of a culturally informed provider training and "dementia friendly clinic" intervention for detection and appropriate management of AI/AN patients with ADRD and MCI in 28 urban and rural clinics serving AI/ANs.

DETAILED DESCRIPTION:
The INTACT team will conduct a group-randomized trial (GRT) to test the effectiveness of the INTACT program, a culturally informed primary care provider training and clinic level workflow intervention for detection and appropriate management of AI/AN patients with Mild Cognitive Impairment (MCI) and ADRD in 28 urban and rural clinics serving AI/ANs. The clinics are the primary unit of randomization. Within each participating clinic, PCPs who are routinely seeing AI/AN patients ages 55 years and older will be recruited for data collection at baseline and 1-year follow-up. Each clinic will be randomized either to the immediate intervention or to a wait-list control arm. Data will be collected from PCP questionnaires, Electronic Health Records (EHR) data extraction and manual medical chart reviews. At the clinic level, we will rely on EHRs to document INTACT's effect on new ADRD diagnoses. At the PCP level, we will test whether INTACT increases knowledge and confidence in dementia assessment, ADRD care, and caregiver support. Patient-level data will be collected from the EHR and by manual chart review.

Once enrolled, clinics will complete a clinic profile interview and clinic and patient population information form, PCPs will be consented and complete a baseline survey. Next the clinics will be randomized into the immediate intervention or the wait-list control arms. Data collection will be conducted at baseline and 1-year follow-up. After completing the 1-year study period, clinics in the wait-list arm will have the opportunity to receive the INTACT intervention.

ELIGIBILITY:
CLINIC Eligibility criteria

To be eligible to participate in INTACT a clinic must be:

1. A primary care clinic
2. Have at least 20 AI/AN active patients 55 years or older
3. Have an EHR system
4. Not intending to change EHR systems in the next year
5. Willing to conduct a total of 40 limited patient chart reviews to assess quality of care metrics for AI/AN patients with MCI and ADRD, staff permitting

PCP

Eligibility criteria:

To be eligible to participate in the baseline and follow-up surveys a primary care provider must be:

1. have a title of MD, DO, Nurse Practitioner, or PA, and
2. regularly provides care to AI/ANs aged 65 and older.

PATIENTS

We will only collect patient EHR data from eligible patients who:

1. Recorded as AI/AN in the EHR system
2. Active clinic patient with prevalent ADRD as of the first day of the time period each data extraction will cover
3. Age 55 or older at the start of the surveillance interval
4. At least one primary care clinic visit during the time period each data extraction will cover.

There are no exclusion criteria for the clinic, PCPs and patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinic Level - new diagnoses of ADRD and MCI (Aim 2) | Baseline and 12-month follow-up
  Primary outcome (as obtained directly from EHRs) will reflect the aggregate counts of new diagnoses (MCI, ADRD, other dementia) during the study period, based on the ICD-10 codes for these diagnoses.
PCP level - care confidence (Aim 1) | Baseline and a 12-month follow-up
  Within each clinic, each participating PCP will complete a baseline and a 12-month follow-up survey. The PCP level primary outcome is care confidence in providing dementia care to patients and their families. Care confience wil be measured using the General Practitioners Confidence and Attitude scale for Dementia (GPACS-D) whic uses a 5 point Likert scale from 1 (strongly agree) to 5 (strongly disagree). The GPACS-D scale has 3 subscales:
  1. Confidence in Clinical Abilities for which a lower score means a better outcome
  2. Attitude to Care for which a lower score means a better outcome
  3. Engagement for which a higher score means a better outcome
Patient level - quality of care 1 (Aim 3) | Baseline and a 12-month follow-up
  Primary outcome (as obtained directly from EHRs) will reflect the number and type of ADRD diagnostic tests.
Patient level - quality of care 2 (Aim 3) | Baseline and a 12-month follow-up
  Primary outcome (as obtained directly from EHRs) will reflect the number of prescriptions of appropriate medications for cognitive and mood symptoms.
Patient level - quality of care 3 (Aim 3) | Baseline and a 12-month follow-up
  Primary outcome (as obtained directly from EHRs) will reflect the number of annual cognitive assessments.
Patient level - quality of care 4 (Aim 3) | Baseline and a 12-month follow-up
  Primary outcome (as obtained directly from EHRs) will reflect the number advance care directive.
Patient level - quality of care 5 (Aim 3) | Baseline and a 12-month follow-up
  Primary outcome (as obtained directly from EHRs) will reflect the number of annual evauations of functional status.
Patient level - quality of care 5 (Aim 3) | Baseline and a 12-month follow-up
  Primary outcome (as obtained directly from EHRs) will reflect the number of pharmacoligical treatment changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT06397339/Prot_SAP_000.pdf